CLINICAL TRIAL: NCT00512551
Title: A Pilot Study of Early Changes in DNA Array Expression Following Chemo-Radiation Treatment of Cervical Cancer
Brief Title: DNA Array Analysis of Patients With Cervical Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: IDP00-075
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; DNA Array Analysis; Gene Expression; DNA
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two biopsies of the cervix will be performed to obtain tumor cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cervical cancer tumor biopsy + radiation therapy: Cervical cancer tumor biopsy + radiation therapy.
  Interventions: Procedure: Tumor Biopsies

INTERVENTIONS:
Procedure: Tumor Biopsies — Biopsies of the cervical tumor performed first before any treatment is given, and the second about 48 hours after radiation treatment has began.

SUMMARY:
The goal of this clinical research study is to find out if the expression of certain genes is linked with the response of cervical cancer to radiation. Researchers will study a large number of genes located in tumor material to learn this information.

DETAILED DESCRIPTION:
Patients in this study are already scheduled to begin radiation therapy. Researchers will get tumor cells by taking two biopsies of the cervix. The first biopsy of the cervical tumor will be done before any treatment is given. The second biopsy will be performed about 48 hours after the radiation treatment has begun. They will then study the cells in the lab with a new technique for studying gene expression called DNA array, as well as human papillomavirus (HPV) analysis, quantification of apoptosis levels, hematoxylin and eosin staining, and storage of tissue for future research.

The patterns of gene expression in the biopsies will be compared with the success of radiation treatments.

Some of the material will also be stored and used in the future for other research projects.

This is an investigational study. A total of 18 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed cervical cancer: clinical Stage IB -IIIB
2. Invasive pure squamous cell carcinoma
3. Planned treatment with concurrent cisplatinum/5-fluorouracil chemotherapy and pelvic radiation

Exclusion Criteria:

1. Previous cervical cancer treatment including but not limited to transvaginal cone irradiation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cervical cancer already scheduled to begin radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2000-06-20 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
The goal of this clinical research study is to find out if the expression of certain genes is linked with the response of cervical cancer to radiation. | 8 Years

SECONDARY OUTCOMES:
Researchers will study a large number of genes located in tumor material to learn this information. | 8 Years

CONTACTS AND LOCATIONS:
Overall Officials: Anuja Jhingran, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org